CLINICAL TRIAL: NCT02869087
Title: DESappear Study: Drug Eluting Scaffold With an Absorbable Platform for Primary Lower Extremity Arterial Revascularization
Brief Title: The DESappear Study: Drug Eluting Scaffold
Acronym: DESappear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Collaborators: Syntactx (Network); Massachusetts General Hospital (Other); Genae (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX CL 1501
Record Dates: First submitted 2016-05-31; First posted 2016-08-16 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental): Single Arm study, study subjects are assigned to treatment with the Akesys Prava Scaffold
  Interventions: Device: Akesys Prava Scaffold

INTERVENTIONS:
Device: Akesys Prava Scaffold — Implantation of the Akesys Prava Sirolimus Eluting Bioresorbable Peripheral Scaffold System

SUMMARY:
The aim of this study is to prospectively collect information to evaluate the safety and performance of the Akesys Prava Sirolimus Eluting Bioresorbable Peripheral scaffold system for the treatment of symptomatic primary atherosclerotic stenoses and occlusions of the superficial femoral artery (SFA).

DETAILED DESCRIPTION:
This is a mutli center, prospective ,single arm study enrolling up to 60 patients at up to 12 centers in New Zealand and Europe.

The purpose is to prospectively collect information to evaluate the safety and performance of the Akesys Prava Sirolimus eluting bioresorbable scaffold system in peripheral arterial disease (PAD) Patients will be treated with the investigational device and followed up clinically at 1 month, 6 Months, 12 months, 24 months and 36 months post procedure.

Patients will undergo non-invasive assessments such as Duplex Ultrasound (DUS), Ankle/Brachial Index (ABI) measurements and will complete a Walking Impairment Questionnaire (WIQ) and Quality of Life Questionnaire (VASCUQoL) at each follow up interval.

Data will be collected via electronic data capture (EDC) and reportable Events will be reviewed by a medical monitor and classified using the MedDRA system. The information entered by the research centres will be source data verified (monitored) by an independent Contract Research Organisation (CRO.) A Data Monitoring Committee (DMC) with appropriately qualified members independent of the study will meet to review and adjudicate on events at predetermined intervals, according to the charter.

Primary safety and efficacy endpoints will be evaluated at 6 months There will be no formal hypothesis testing in the study, endpoints will be evaluated with 95% confidence intervals around the observed point estimates. The endpoints will be evaluated with Kaplan-Meier methodology.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

1. Subject is ≥18 years of age.
2. Subject has been informed of the nature of the study, agrees to its provisions, is able to provide informed consent, and agrees to undergo all protocol-required follow up examinations and requirements.
3. Subject's life expectancy is at least 1 year.
4. Subject is diagnosed as having symptomatic claudication (Rutherford-Becker Clinical Category 2-4).
5. For females of childbearing potential, a negative pregnancy test within 14 days before index procedure is required
6. Subject is able to take a P2Y12 receptor antagonist (e.g. clopidogrel, ticagrelor, prasugrel or ticagrelor) and acetylsalicylic acid (aspirin).

Angiographic inclusion criteria:

1. A single, de novo native disease segment of the SFA
2. Proximal margin of target lesion is ≥1 cm distal to the common femoral artery bifurcation; distal margin of target lesion is within the SFA.
3. Vessel diameter from ≥5.0 mm to ≤6.0 mm evaluated by on-line quantitative vascular angiography (QVA) after pre-dilatation per core laboratory guidelines.
4. Target lesion diameter reduction ≥50%
5. Target lesion length ≤53 mm
6. Patent inflow artery free from significant lesion (≥50% diameter reduction;
7. Patent distal popliteal artery free from significant lesion (≥50%) with angiographic demonstration of at least one fully patent distal outflow artery (anterior tibial, posterior tibial, or peroneal) to its terminus.

Exclusion Criteria:

Clinical exclusion criteria:

1. Previous bypass surgery or stenting at the TL;
2. Percutaneous or open surgical revascularization of the contralateral iliac or infrainguinal arteries ≤30 days prior to the planned index procedure. Iliac artery lesions may be treated during the index procedure if necessary for approach to the TL;
3. Failure to successfully cross the target lesion with a guide wire;
4. Subject has a known abdominal aortic aneurysm >4 cm in diameter, a known iliac artery aneurysm >3 cm in diameter, or history of open surgical abdominal aortic or iliac revascularization.
5. Lesion within or adjacent to an aneurysm or presence of a popliteal aneurysm;
6. Subject is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus);
7. Acute limb ischemia;
8. History of a bleeding diathesis;
9. History of a hypercoagulability syndrome;
10. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3; a WBC <3,000 cells/mm3; or hemoglobin <10.0 g/dL;
11. Acute or chronic renal dysfunction (creatinine >2.5 mg/dl or >176 μmol/L), or on chronic hemodialysis;
12. Severe liver impairment as defined by total bilirubin ≥3 mg/dl or two times increase over the normal level of SGOT/AST or SGPT/ALT;
13. Known allergies to the following: aspirin, clopidogrel, prasugrel, ticagrelor, or heparin, contrast agent (that cannot be adequately premedicated), or drugs similar to sirolimus (i.e. tacrolimus, everolimus, zotarolimus) or other macrolides;
14. Subject requires planned procedure within 30 days that would necessitate the discontinuation of clopidogrel, prasugrel, or ticagrelor;
15. Subject is on chronic Coumadin therapy
16. Subject has had or is planned to have treatment with DES or drug coated balloon (DCB) within 90 days pre- or post-index procedure;
17. Subject is non-ambulatory;
18. Subject has undergone percutaneous intervention of the coronary, carotid, or arterial bed exclusive of the <30 days prior to the planned index procedure.
19. Subject has received, or is on the waiting list for, an organ transplant;
20. Subject had a myocardial infarction (MI) within the previous 30 days prior to the planned index procedure;
21. Subject has had a stroke within the previous 30 days of the planned index procedure and/or has deficits from a prior stroke that limit the subject's ability to walk;
22. Subject has unstable angina defined as rest angina with ECG changes;
23. Subject has a groin infection, or an acute systemic infection that has not been treated successfully or is currently under treatment;
24. Subject has acute thrombophlebitis (superficial or deep) in either extremity;
25. Subject has other medical conditions (e.g., cancer, congestive heart failure or substance abuse) that may cause the subject to be non-compliant with protocol requirements or confound data interpretation;
26. Subject is currently participating or wanting to participate in a clinical trial following 6 months after the index procedure in an investigational drug, biologic, or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials);
27. Subject is unable to understand or unwilling to cooperate with study procedures;
28. Subject has prior minor or major amputation of either lower extremity;
29. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give informed consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy;
30. Pre-operative plan for additional treatment of the target lesion at the time of the study procedure with alternative therapy such as drug-eluting stent (DES) and scaffold, laser, atherectomy, cryoplasty, cutting balloon, drug-eluting balloon, or brachytherapy (vessel preparation with uncoated balloon angioplasty is allowed); 31Plan for cardiovascular surgical or interventional procedure ≤30 days after the study procedure including planned treatment of the contralateral lower extremity.

Angiographic exclusion criteria:

1. Target extremity has an angiographically significant (>50% diameter reduction) lesion located in the target vessel distal to the target lesion;
2. Thrombus in the target vessel;
3. Stenosis (>50%) or occlusion of an ipsilateral inflow artery;
4. Angiographic evidence of thromboembolism or atheroembolism from treatment of an ipsilateral iliac lesion, or from crossing or pre-dilating the target lesion;
5. Target lesion has calcification with either of the following characteristics:

   * Circumferential orientation, or
   * Thickness >2 mm (radially) within the wall of the target lesion.
6. Failure to achieve less than 30% residual stenosis after balloon predilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Freedom from composite of perioperative death < 30 days and freedom from major adverse limb events (MALE) defined as the occurrence of major amputation, thrombectomy, thrombolysis or major open surgical revascularization | 6 months
  Primary Safety Endpoint
Primary Patency defined as the freedom from restenosis (>50% diameter reduction defined by Duplex Ultrasound) or clinically driven target lesion revascularization through 6 months | 6 months
  Primary Effectiveness Endpoint

SECONDARY OUTCOMES:
Freedom from composite of perioperative death within 30 days and freedom from major adverse limb events (MALE) defined as the occurrence of major amputation, thrombectomy, thrombolysis or major open surgical revascularization. | 12 months
  Secondary Safety endpoint
Freedom from the composite of target lesion (TL) occlusion, reintervention or restenosis defined as a >50% diameter reduction in the target lesion, as confirmed by Duplex Ultrasound or angiography | 12 months
  Secondary Effectiveness Endpoint
All cause mortality | 12 months
Technical Success defined as the successful delivery and deployment of the device assessed by angiography at the conclusion of the procedure | Post Procedure- Procedure may take up to 2 hours
  The assessment will be made and evaluated at the conclusion of the index procedure
Technical Success defined as no implantation of metallic stent assessed by angiography at the conclusion of the procedure | Post Procedure, procedure may take up to 2 hours
  the assessment will be made and evaluated at the conclusion of the Index procedure
Technical Success defined as < 30%residual stenosis after successful implantation of the scaffold assessed by angiography at the conclusion of the procedure | Post Procedure, procedure may take up to 2 hours
  The assessment will be made and evaluated at the conclusion of the index procedure
Major target extremity amputation | 1 month,6 months,12 months, 24 months, 36 months
Minor target extremity amputation | 1 month,6 months,12 months, 24 months, 36 months
Scaffold Thrombosis | 1 month,6 months,12 months, 24 months, 36 months
Target Lesion binary restenosis by duplex ultrasound Peak Systolic Velocity ratio (PSVR>2.4) | 1 month, 6 months,12 months, 24 months, 36 months
Clinically driven target lesion restenosis defined as any intervention due to worsening symptoms, a fall in ABI or TL restenosis as determined by duplex ultrasound | 1 month,6 months,12 months, 24 months, 36 months
Target extremity revascularisation | 1 month,6 months,12 months, 24 months, 36 months
Primary patency of the target lesion | 1 month,6 months,12 months, 24 months, 36 months
Primary assisted patency of the target lesion | 1 month,6 months,12 months, 24 months, 36 months
Secondary patency of the target lesion | 1 month,6 months,12 months, 24 months, 36 months
Rutherford Becker clinical category | 1 month,6 months,12 months, 24 months, 36 months
Ankle Brachial Index in the target extremity | 1 month,6 months,12 months, 24 months, 36 months
Walking Capacity as demonstrated by the Walking Impairment Questionnaire | 1 month,6 months,12 months, 24 months, 36 months
Quality of Life measures using VASCUQoL- disease specific | 1 month,6 months,12 months, 24 months, 36 months
Duplex ultrasound derived Peak Velocity (PSV) at the target lesion | 1 month,6 months,12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, Doctor, Principal Investigator — AZ Sint-Blasius Dendermonde; Dierk Scheinert, Doctor, Principal Investigator — Universitätsklinikum Leipzig
Locations (11):
- Austria (2):
  - LKH University Hospital Graz, Graz, Styria
  - Hanusch Hospital, Vienna
- Belgium (2):
  - AZ Sint Blasius, Dendermonde, Dendermonde, Brussels Capital
  - Heilig Hart Hospital, Tienen
- Germany (5):
  - Bonifatius Hospital, Lingen, Lower Saxony
  - Klinikum Arnsberg, Arnsberg, North Rhine-Westphalia
  - Heart Center Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Leipzig AöR,, Leipzig
  - St Franziskus Hospital, Münster
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No